CLINICAL TRIAL: NCT06286813
Title: The Effect of Almond and Extra Virgin Olive Oils on Maintaining Skin Integrity in Neonates Admitted to the Neonatal Intensive Care Unit
Brief Title: The Effect of Almond and Extra Virgin Olive Oils on Maintaining Skin Integrity in Neonates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Akarakoc
Record Dates: First submitted 2024-02-09; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Skin Care
Keywords: Newborn, skin care, extra virgin olive oil, almond oil.
MeSH Terms: interventions — Oils

STUDY DESIGN:
Intervention Model Description: Interventional research with two parallel groups (almond olive group and virgin olive oil group) and no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond oil group (Experimental): On the first day of neonates' admission to the clinic, their skin condition will be evaluated using the NSCS, and the hydration of skin will be measured using a digital moisture meter with the recommended usage guide. During morning care at 09:00 a.m., almond oil (10 ml) will be applied to their entire body, except for the head. Three hours after the application, at 12:00 a.m., their skin condition will be assessed, and the hydration will be measured and recorded. This application will continue for 5 days.
  Interventions: Other: Plant (natural) oils
- Extra Virgin Olive Oil Group (Experimental): On the first day of neonates' admission to the clinic, their skin condition will be evaluated using the NSCS, and the hydration of skin will be measured using a digital moisture meter with the recommended usage guide. During morning care at 09:00 a.m., extra virgin olive oil(10 ml) will be applied to their entire body, except for the head. Three hours after the application, at 12:00 a.m., their skin condition will be assessed, and the hydration will be measured and recorded. This application will continue for 5 days.
  Interventions: Other: Plant (natural) oils

INTERVENTIONS:
Other: Plant (natural) oils — Using 10 ml of plant(natural) oil once a day for daily skin care of newborns

SUMMARY:
This study aimed to evaluate the effects of extra virgin olive and almond oils on maintaining skin integrity in neonates admitted to the neonatal intensive care unit.

Interventional research with two parallel groups and no control group

DETAILED DESCRIPTION:
The study was conducted in the Neonatal intensive care unit (NICU) of a training and research hospital.The total number of infants admitted to the NICU was 28. Each nurse is responsible for the care of 3 or 4 newborn babies.

Skin are routines in the NICU: A skin condition assessment score is routinely performed every day (09.00 am) in all infants and moisturizing products are used for their skin care. Therefore, there was no control group in the study.

Extra virgin olive oil and almond oil are among the skin care products used in the clinic routines. Therefore, the effects of the currently used oils were compared in the study

ELIGIBILITY:
Inclusion Criteria:

* Neonates who were born at 37-42 weeks of gestation, were planned to be hospitalized in the NICU for at least 5 days, had a post-natal age of 0-72 hours, and were received written and verbal consent from parents were included in the study.

Exclusion Criteria:

* ; Neonates who were discharged before 5 days and required phototherapy were excluded from the study.

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-03-02 (Estimated); Primary Completion 2024-05-03 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Neonatal skin condition score | 5 days
  This is a three-point Likert-type scale to evaluate dryness, redness, peeling / deterioration in newborn baby skin. For each criterion in the evaluation of the scale score; 1 refers to the best and 3 to the worst skin condition. The highest and lowest scores on the scale are 9 and 3, respectively. A higher scale score indicates poorer skin condition
Skin moisture meter(DMM): | 5 days
  The product shows the moisture level (0%-99.9%) in contact with the skin and does not harm the skin. It provides measurement results with high precision

CONTACTS AND LOCATIONS:
Overall Officials: AYŞE KARAKOÇ, Study Director — Marmara University
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Title of study and method
Supporting Information: Study Protocol
Time Frame: starting 3 months after publication
Access Criteria: with e-mail (akarakoc@marmara.edu.tr)

REFERENCES:
- [Derived] Topcuoglu Arslan IZ, Karakoc A. Effect of Almond and Extra Virgin Olive Oils on Maintaining Skin Integrity in Neonates Admitted to the Neonatal Intensive Care Unit. Adv Skin Wound Care. 2025 Aug 1;38(7):381-386. doi: 10.1097/ASW.0000000000000306. Epub 2025 Apr 4. PMID 40184517